CLINICAL TRIAL: NCT04116749
Title: Comparison of Gastric Emptying of Water in Obese vs. Non-obese Term Pregnant Women Undergoing Elective Cesarean Section
Brief Title: Gastric Emptying of Water in Obese Term Pregnant Women
Status: Terminated | Type: Observational
Why Stopped: Unavailable to collect study participants.
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Eunah Cho, MD, Clinical Assistant Professor, Kangbuk Samsung Hospital
Other Study IDs: KBSMC 2019-08-039
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Water

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-obese women: body mass index lower than 30 (kg/m^2) at term
  Interventions: Other: Water
- Obese women: body mass index equal or greater than 30 (kg/m^2) at term
  Interventions: Other: Water

INTERVENTIONS:
Other: Water — Drink water freely until 2 hours before anesthesia.

SUMMARY:
It has been believed that the risk of pulmonary aspiration in term pregnant women is increased, and should be considered that all term pregnant women to have "full stomach". Recently, gastric ultrasound has been adopted as a useful tool for quantitative and qualitative assessment of stomach before anesthesia, and predict the risk of pulmonary aspiration.

Although, both the obesity and pregnancy are known to be the risk of pulmonary aspiration, it is suggested in the American Society of Anesthesiology fasting guidelines, that the same fasting time should be applied in the obese and non-obese parturients. However, this was based on one study done in a small (10) numbers of volunteers.

Therefore, the investigators aimed to compare the gastric antral cross-sectional area in both obese and non-obese term pregnant women, scheduled for elective cesarean section.

DETAILED DESCRIPTION:
This study is a prospective, observational study. 42 term (≥37 weeks) pregnant, non-laboring adult women scheduled for cesarean delivery will be included in the study. They will be allowed to drink water freely, until 2 hours before the anesthesia. Gastric ultrasound will be performed in 21 non-obese women, and 21 obese women. The obesity is defined by the body mass index at term.

ELIGIBILITY:
Inclusion Criteria:

* Non laboring, term (≥37 weeks) pregnant women
* Scheduled for elective cesarean section
* aged ≥ 18 years old
* American Society of Anesthesiology physical class 1-3

Exclusion Criteria:

* multigestational pregnancy
* diagnosed for delayed gastric emptying (GERD, gastrointestinal disease)
* diabetes

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing elective cesarean section.
Study Population: Non laboring, term (≥37 weeks) pregnant women uldergoing elective cesarean section, in our medical center.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Gastric antral cross-sectional area | 2 hours after the time allowed to drink water.
  Cross-sectional area of gastric antrum assessed by ultrasonography

SECONDARY OUTCOMES:
Preoperative anxiety | 2 hours after the time allowed to drink water.
  Preoperative anxiety is scored from 0 (never) to 10 (very much).
Hunger score | 2 hours after the time allowed to drink water.
  Hunger score is scored from 0 (never) to 10 (very much).
Thirst score | 2 hours after the time allowed to drink water.
  Thirst score is scored from 0 (never) to 10 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Eunah Cho, MD, Principal Investigator — KangbukSamsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided